CLINICAL TRIAL: NCT05716828
Title: Effect of Balint Group on Burnout and Self-efficacy of Nurse Leaders in China: A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Qu Shan, Head of the Department of Medical Psychology, Peking University People's Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: balint2022
Record Dates: First submitted 2023-01-17; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Burnout; Self Efficacy
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balint group (Experimental): Participants in the Balint group completed Balint training for a period of three months.
  Interventions: Other: Balint group activities
- non-Balint group (No Intervention)

INTERVENTIONS:
Other: Balint group activities — A Balint group is a working form that focuses on the professional doctor-patient relationship. Participants in the Balint group completed Balint training for a period of at least three months, which included two lectures and 10 small group discussion sessions held once a month for one hour at a time (on Thursdays from 12 to 1 PM). Balint group is a closed group including one to two group leaders and six to twelve participants, with sessions lasting 60 to 90 minutes.
  Arms: Balint group

SUMMARY:
Background: Burnout is common among nurses and is related to negative outcomes of medical care. This study aimed to explore the effectiveness of Balint group activities in burnout reduction among nurse leaders in a Chinese hospital.

Methods: This was a randomised controlled trial with a pre- and post-test. A total of 80 nurse leaders were randomly assigned to either a Balint group (n=40) or a non-Balint group (n=40). Participants in the Balint group completed Balint training for a period of three months. Participants in both groups completed the Maslach Burnout Inventory-Human Services Survey (MBI) and the General Self-Efficacy Scale (GSES) at the beginning and end of the study（three months later ）. Balint group members also completed the Group Climate Questionnaire-Short Format the end of the study（three months later ）.

ELIGIBILITY:
Inclusion Criteria:

1. nurse leaders in clinical departments
2. voluntary participation

Exclusion Criteria:

a. previous participation in Balint groups

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Maslach Burnout Inventory-Human Services Survey (MBI-HSS) subscale emotional exhaustion (MBI-EE) | The first time for participants in both groups was assessed the MBI-EE questionnaire at baseline.
  Maslach Burnout Inventory-Human Services Survey (MBI-HSS) includes 22 items across three domains: emotional exhaustion (EE; 9 items), depersonalization (DP; 5 items), and personal accomplishment (PA; 8 items). The scoring range for each item is 0 (never felt) to 6 (felt every day). The EE subscale evaluates the feeling of excessive emotional stress and exhaustion due to work, which is characterized by mental, emotional, and physical exhaustion
Maslach Burnout Inventory-Human Services Survey (MBI-HSS) subscale emotional exhaustion (MBI-EE) | The second time for participants in both groups was assessed the MBI-EE questionnaire through Balint group activities completion, 3 months later
  Maslach Burnout Inventory-Human Services Survey (MBI-HSS) includes 22 items across three domains: emotional exhaustion (EE; 9 items), depersonalization (DP; 5 items), and personal accomplishment (PA; 8 items). The scoring range for each item is 0 (never felt) to 6 (felt every day). The EE subscale evaluates the feeling of excessive emotional stress and exhaustion due to work, which is characterized by mental, emotional, and physical exhaustion
Maslach Burnout Inventory-Human Services Survey (MBI-HSS) subscale depersonalization (MBI-DP) | The first time for participants in both groups was assessed the MBI-DP questionnaire at baseline.
  Maslach Burnout Inventory-Human Services Survey (MBI-HSS) includes 22 items across three domains: emotional exhaustion (EE; 9 items), depersonalization (DP; 5 items), and personal accomplishment (PA; 8 items). The scoring range for each item is 0 (never felt) to 6 (felt every day). The DP subscale measures unsympathetic and impersonal response to patients, and is regarded as a form of alienation.
Maslach Burnout Inventory-Human Services Survey (MBI-HSS) subscale depersonalization (MBI-DP) | The second time for participants in both groups was assessed the MBI-DP questionnaire through Balint group activities completion, 3 months later
  Maslach Burnout Inventory-Human Services Survey (MBI-HSS) includes 22 items across three domains: emotional exhaustion (EE; 9 items), depersonalization (DP; 5 items), and personal accomplishment (PA; 8 items). The scoring range for each item is 0 (never felt) to 6 (felt every day). The DP subscale measures unsympathetic and impersonal response to patients, and is regarded as a form of alienation.
Maslach Burnout Inventory-Human Services Survey (MBI-HSS) subscale personal accomplishment (MBI- PA) | The first time for participants in both groups was assessed the MBI-PA questionnaire at baseline.
  Maslach Burnout Inventory-Human Services Survey (MBI-HSS) includes 22 items across three domains: emotional exhaustion (EE; 9 items), depersonalization (DP; 5 items), and personal accomplishment (PA; 8 items). The scoring range for each item is 0 (never felt) to 6 (felt every day). The PA subscale assesses work-related ability and sense of accomplishment .
Maslach Burnout Inventory-Human Services Survey (MBI-HSS) subscale personal accomplishment (MBI- PA) | The second time for participants in both groups was assessed the MBI-PA questionnaire through Balint group activities completion, 3 months later
  Maslach Burnout Inventory-Human Services Survey (MBI-HSS) includes 22 items across three domains: emotional exhaustion (EE; 9 items), depersonalization (DP; 5 items), and personal accomplishment (PA; 8 items). The scoring range for each item is 0 (never felt) to 6 (felt every day). The PA subscale assesses work-related ability and sense of accomplishment .

SECONDARY OUTCOMES:
The General Self-Efficacy Scale (GSES) | The first time for participants in both groups was assessed the GSES questionnaire at baseline.
  The General Self-Efficacy Scale (GSES) is a 10-item scale used to measure individuals' overall self-confidence in dealing with different environmental challenges or unprecedented situations. Participants are asked to rate 10 questions by choosing one of four response options: 1 (completely incorrect), 2 (almost incorrect), 3 (relatively correct), or 4 (completely correct). A higher score indicates a higher level of general self-efficacy.
The General Self-Efficacy Scale (GSES) | The second time for participants in both groups was assessed the GSES questionnaire through Balint group activities completion, 3 months later
  The General Self-Efficacy Scale (GSES) is a 10-item scale used to measure individuals' overall self-confidence in dealing with different environmental challenges or unprecedented situations. Participants are asked to rate 10 questions by choosing one of four response options: 1 (completely incorrect), 2 (almost incorrect), 3 (relatively correct), or 4 (completely correct). A higher score indicates a higher level of general self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Shan Qu, Qu, Principal Investigator — Peking University People's Hospital
Locations (1):
- Shan Qu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Minjie Z, Zhijuan X, Xinxin S, Xinzhu B, Shan Q. The effects of cognitive behavioral therapy on health-related quality of life, anxiety, depression, illness perception, and in atrial fibrillation patients: a six-month longitudinal study. BMC Psychol. 2023 Dec 7;11(1):431. doi: 10.1186/s40359-023-01457-z. PMID 38062475